CLINICAL TRIAL: NCT03563157
Title: NANT Colorectal Cancer (CRC) Vaccine: A Phase 1b/2 Trial of the NANT CRC Vaccine vs Regorafenib in Subjects With Metastatic CRC Who Have Been Previously Treated With Standard-of-Care Therapy
Brief Title: QUILT 3.071: NANT Colorectal Cancer (CRC) Vaccine
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: low enrollment
Sponsor: ImmunityBio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: QUILT-3.071
Record Dates: First submitted 2018-05-22; First posted 2018-06-20 (Actual); Results first posted 2024-12-11 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Colorectal Cancer Metastatic; mCRC
Keywords: Colorectal Cancer; Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — ALT-803; yeast-CEA vaccine; avelumab; Capecitabine; Cetuximab; Cyclophosphamide; Fluorouracil; Leucovorin; 130-nm albumin-bound paclitaxel; Oxaliplatin; regorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- NANT Colorectal Cancer (CRC) Vaccine (Experimental): A combination of agents will be administered to subjects in this study: Aldoxorubicin HCI, ETBX-011, ETBX-021, ETBX-051, ETBX-061, GI-4000, GI-6207, GI-6301, haNK, N-803, Avelumab, Capecitabine, Cetuximab, Cyclophosphamide, 5-Fluorouracil, Leucovorin, Nab-paclitaxel, Oxaliplatin, Regorafenib, SBRT.
  Interventions: Biological: Aldoxorubicin Hydrochloride; Biological: ALT-803; Biological: ETBX-011; Biological: ETBX-021; Biological: ETBX-051; Biological: ETBX-061; Biological: GI-4000; Biological: GI-6207; Biological: GI-6301; Biological: haNK; Drug: Avelumab; Drug: Capecitabine; Drug: Cetuximab; Drug: Cyclophosphamide; Drug: 5-Fluorouracil; Drug: Leucovorin; Drug: Nab-paclitaxel; Drug: Oxaliplatin; Drug: Regorafenib; Procedure: SBRT
- Regorafenib (Active Comparator): Regorafenib will be administered to subjects in this study.
  Interventions: Drug: Regorafenib

INTERVENTIONS:
Biological: Aldoxorubicin Hydrochloride — Aldoxorubicin Hydrochloride HCI
  Arms: NANT Colorectal Cancer (CRC) Vaccine
Biological: ALT-803 — Recombinant human super agonist interleukin-15 (IL-15) complex [also known as IL-15N72D;IL-15RaSu/IgG1 Fe complex1]
  Arms: NANT Colorectal Cancer (CRC) Vaccine
Biological: ETBX-011 — Ad5 [E1-, E2b-]-CEA
  Arms: NANT Colorectal Cancer (CRC) Vaccine
Biological: ETBX-021 — Ad5 [E1-, E2b-]-[HER2]
  Arms: NANT Colorectal Cancer (CRC) Vaccine
Biological: ETBX-051 — Ad5 [E1-, E2b-]-Brachyury
  Arms: NANT Colorectal Cancer (CRC) Vaccine
Biological: ETBX-061 — Ad5 [E1-, E2b-]-mucin 1 [MUC1]
  Arms: NANT Colorectal Cancer (CRC) Vaccine
Biological: GI-4000 — RAS yeast
  Arms: NANT Colorectal Cancer (CRC) Vaccine
Biological: GI-6207 — CEA yeast
  Arms: NANT Colorectal Cancer (CRC) Vaccine
Biological: GI-6301 — Brachyury yeast
  Arms: NANT Colorectal Cancer (CRC) Vaccine
Biological: haNK — haNK™, NK-92 [CD16.158V, ER IL-2]
  Arms: NANT Colorectal Cancer (CRC) Vaccine
Drug: Avelumab — BAVENCIO® injection
  Arms: NANT Colorectal Cancer (CRC) Vaccine
Drug: Capecitabine — XELODA® tablets
  Arms: NANT Colorectal Cancer (CRC) Vaccine
Drug: Cetuximab — ERBITUX® injection
  Arms: NANT Colorectal Cancer (CRC) Vaccine
Drug: Cyclophosphamide — Cyclophosphamide Capsules
  Arms: NANT Colorectal Cancer (CRC) Vaccine
Drug: 5-Fluorouracil — 5-FU; Fluorouracil Injection
  Arms: NANT Colorectal Cancer (CRC) Vaccine
Drug: Leucovorin — Leucovorin Calcium
  Arms: NANT Colorectal Cancer (CRC) Vaccine
Drug: Nab-paclitaxel — ABRAXANE® for Injectable Suspension [paclitaxel protein-bound particles for injectable suspension] [albumin-bound]
  Arms: NANT Colorectal Cancer (CRC) Vaccine
Drug: Oxaliplatin — ELOXATIN® injection
  Arms: NANT Colorectal Cancer (CRC) Vaccine
Drug: Regorafenib — STIVARGA® tablets
Procedure: SBRT — Stereotactic body radiation therapy
  Arms: NANT Colorectal Cancer (CRC) Vaccine

SUMMARY:
QUILT 3.071 NANT Colorectal Cancer (CRC) Vaccine: This is a Phase 1b/2 study investigating the effect of NANT CRC vaccine vs regorafenib in subjects with CRC who were previously treated with SOC.

DETAILED DESCRIPTION:
NANT Colorectal Cancer (CRC) Vaccine: A phase 1b/2 Trial of the NANT CRC Vaccine vs Regorafenib in Subjects with Metastatic CRC Who Have Been Previously Treated with Standard-Of-Care Therapy

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. Able to understand and provide a signed informed consent that fulfills the relevant IRB or IEC guidelines.
3. Histologically-confirmed recurrent or metastatic CRC previously treated with fluoropyrimidine-, oxaliplatin- and irinotecan-based chemotherapy, an anti-VEGF biological therapy, and if RAS wild-type, an anti-EGFR therapy; or subjects who are ineligible for these therapies.
4. ECOG performance status of 0 or 1.
5. Have at least 1 measurable lesion of ≥ 1.0 cm.
6. Must have a recent FFPE tumor biopsy specimen following the conclusion of the most recent anticancer treatment and be willing to release the specimen for prospective and exploratory tumor molecular profiling. If an historic specimen is not available, the subject must be willing to undergo a biopsy during the screening period, if considered safe by the Investigator. If safety concerns preclude collection of a biopsy during the screening period, a tumor biopsy specimen collected prior to the conclusion of the most recent anticancer treatment may be used.
7. Must be willing to provide blood samples prior to the start of treatment on this study for prospective tumor molecular profiling and exploratory analyses.
8. Must be willing to provide a tumor biopsy specimen 8 weeks after the start of treatment for exploratory analyses, if considered safe by the Investigator.
9. Ability to attend required study visits and return for adequate follow-up, as required by this protocol.
10. Agreement to practice effective contraception for female subjects of child-bearing potential and non-sterile males. Female subjects of child-bearing potential must agree to use effective contraception for up to 1 year after completion of therapy, and non- sterile male subjects must agree to use a condom for up to 4 months after treatment. Effective contraception includes surgical sterilization (eg, vasectomy, tubal ligation), two forms of barrier methods (eg, condom, diaphragm) used with spermicide, IUDs, and abstinence.

    Phase 2 single-arm component only
11. Must have progressed on or after regorafenib treatment in the randomized phase 2 portion of the study OR progressed or experienced unacceptable toxicity on SoC and regorafenib prior to enrollment on the study.

Exclusion Criteria:

1. MSI-high or MMR-deficient tumors eligible for, but not yet treated with, a PD-1 inhibitor.
2. Serious uncontrolled concomitant disease that would contraindicate the use of the investigational drugs used in this study or that would put the subject at high risk for treatment-related complications.
3. Systemic autoimmune disease (eg, lupus erythematosus, rheumatoid arthritis, Addison's disease, or autoimmune disease associated with lymphoma).
4. History of organ transplant requiring immunosuppression.
5. History of or active inflammatory bowel disease (eg, Crohn's disease, ulcerative colitis).
6. Inadequate organ function, evidenced by the following laboratory results:

   1. ANC < 1,000 cells/mm^3.
   2. Uncorrectable grade 3 anemia (hemoglobin < 8 g/dL)
   3. Platelet count < 75,000 cells/mm^3.
   4. Total bilirubin > ULN (unless the subject has documented Gilbert's syndrome).
   5. AST (SGOT) or ALT (SGPT) > 2.5 × ULN (> 5 × ULN in subjects with liver metastases).
   6. ALP > 2.5 × ULN (> 5 × ULN in subjects with liver metastases, or >10 × ULN in subjects with bone metastases).
   7. Serum creatinine > 2.0 mg/dL or 177 μmol/L.
   8. Serum anion gap > 16 mEq/L or arterial blood with pH < 7.3.
7. Uncontrolled hypertension (systolic > 160 mm Hg and/or diastolic > 110 mm Hg) or clinically significant (ie, active) cardiovascular disease, cerebrovascular accident/stroke, or myocardial infarction within 6 months prior to first study medication; unstable angina; congestive heart failure of New York Heart Association grade 2 or higher; or serious cardiac arrhythmia requiring medication. Subjects with uncontrolled hypertension should be medically managed on a stable regimen to control hypertension prior to study entry.
8. Serious myocardial dysfunction defined by ECHO as absolute LVEF 10% below the institution's lower limit of predicted normal.
9. Dyspnea at rest due to complications of advanced malignancy or other disease requiring continuous oxygen therapy.
10. Positive results of screening test for HIV.
11. Current chronic daily treatment (continuous for > 3 months) with systemic corticosteroids (dose equivalent to or greater than 10 mg/day methylprednisolone), excluding inhaled steroids. Short-term steroid use to prevent IV contrast allergic reaction or anaphylaxis in subjects who have known contrast allergies is allowed.
12. Known hypersensitivity to any component of the study medication(s).
13. Subjects taking any medication(s) (herbal or prescribed) known to have an adverse drug reaction with any of the study medications.
14. Concurrent or prior use of a strong CYP3A4 inhibitor (including ketoconazole, itraconazole, posaconazole, clarithromycin, indinavir, nefazodone, nelfinavir, ritonavir, saquinavir, telithromycin, voriconazole, and grapefruit products) or strong CYP3A4 inducers (including phenytoin, carbamazepine, rifampin, rifabutin, rifapentin, phenobarbital, and St John's Wort) within 14 days before study day 1.
15. Concurrent or prior use of a strong CYP2C8 inhibitor (gemfibrozil) or moderate CYP2C8 inducer (rifampin) within 14 days before study day 1.
16. Participation in an investigational drug study or history of receiving any investigational treatment within 30 days prior to screening for this study, except for testosterone-lowering therapy in men with prostate cancer.
17. Assessed by the Investigator to be unable or unwilling to comply with the requirements of the protocol.
18. Concurrent participation in any interventional clinical trial.
19. Pregnant and nursing women.

    Phase 2 randomized component only
20. Prior regorafenib treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2018-09-28 (Actual); Primary Completion 2019-04-21 (Actual); Study Completion 2019-08-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Chan Soon-Shiong Institute for Medicine, El Segundo, California, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Only the Phase 1b portion of the study enrolled participants. The study was terminated early, so no participants were enrolled on the Phase 2 portion of the study.
  Eligible participants could have gone through both induction and maintenance treatment on study.
  All subjects were treated on the same arm and not randomized in the Phase 1b portion of the study.
Groups:
- NANT Colorectal Cancer (CRC) Vaccine: A combination of agents was administered to subjects in this study: Aldoxorubicin HCI, ETBX-011, ETBX-021, ETBX-051, ETBX-061, GI-4000, GI-6207, GI-6301, haNK, N-803, Avelumab, Capecitabine, Cetuximab, Cyclophosphamide, 5-Fluorouracil, Leucovorin, Nab-paclitaxel, Oxaliplatin, Regorafenib, SBRT.
  Aldoxorubicin Hydrochloride: Aldoxorubicin Hydrochloride HCI
  ALT-803: Recombinant human super agonist interleukin-15 (IL-15) complex [also known as IL-15N72D;IL-15RaSu/IgG1 Fe complex1]
  ETBX-011: Ad5 [E1-, E2b-]-CEA
  ETBX-021: Ad5 [E1-, E2b-]-[HER2]
  ETBX-051: Ad5 [E1-, E2b-]-Brachyury
  ETBX-061: Ad5 [E1-, E2b-]-mucin 1 [MUC1]
  GI-4000: RAS yeast
  GI-6207: CEA yeast
  GI-6301: Brachyury yeast
  haNK: haNK™, NK-92 [CD16.158V, ER IL-2]
  Avelumab: BAVENCIO® injection
  Capecitabine: XELODA® tablets
  Cetuximab: ERBITUX® injection
  Cyclophosphamide: Cyclophosphamide Capsules
  5-Fluorouracil: 5-FU; Fluorouracil Injection
  Leucovorin: Leucovorin Calcium
  Nab-paclitaxel: ABRAXANE® for Injectable Suspension [paclitaxel protein-bound particles for injectable suspension] [albumin-bound]
  Oxaliplatin: ELOXATIN® injection
  Regorafenib: STIVARGA® tablets
  SBRT: Stereotactic body radiation therapy
Period: Overall Study
Arm/Group | NANT Colorectal Cancer (CRC) Vaccine
Started | 2
Completed | 0
Not Completed | 2
Not completed — Progressive Disease | 2

BASELINE CHARACTERISTICS:
Arm/Group | NANT Colorectal Cancer (CRC) Vaccine
Number analyzed (Participants) | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.0 (4.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 1
SUBJECTS WITH METASTATIC CRC WHO HAVE BEEN PREVIOUSLY TREATED WITH STANDARD-OF-CARE (SOC) THERAPY [Count of Participants; unit: Participants] | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (AEs) and Serious AEs (SAEs)
Description: Graded Using the National Cancer Institute(NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 4.03
Time Frame: 30 days after last dose, up to 6 months or until they experience confirmed progressive disease or unacceptable toxicity, withdrawn consent, or if the Investigator feels it is no longer in their best interest.
Measure: Count of Participants; unit: Participants
Arm/Group | NANT Colorectal Cancer (CRC) Vaccine
Number analyzed (Participants) | 2
Participants
  Treatment Emergent Adverse Events | 2
  Treatment Emergent Serious Adverse Events | 1

2. Secondary Outcome: Objective Response Rate by RECIST Version 1.1 and irRC
Description: Tumors were assessed at screening, and tumor response will be assessed every 8 weeks during the induction phase, and every 12 weeks during the maintenance phase by computed tomography (CT) or magnetic resonance imaging (MRI) of target and non-target lesions in accordance with RECIST Version 1.1.
  An objective response is defined as a confirmed complete or partial overall response with confirmation occurring at least 4 weeks after the initial response is observed.
Time Frame: Tumors were assessed at screening, and tumor response will be assessed every 8 weeks during the induction phase, and every 12 weeks during the maintenance phase until disease progression, up to 4 months
Measure: Count of Participants; unit: Participants
Arm/Group | NANT Colorectal Cancer (CRC) Vaccine
Number analyzed (Participants) | 2
Participants | 0

3. Secondary Outcome: Progression Free Survival by RECIST Version 1.1 and irRC
Description: PFS was evaluated using Kaplan-Meier methods. PFS was defined as the time from the date of first treatment to the date of disease progression or death (any cause) whichever occurs first. Subjects completing study follow-up or initiating a new anticancer therapy prior to documented PD was censored in the PFS analysis at the last known date the subject was progression free prior to completing follow-up or initiating the new therapy.
Time Frame: Tumors were assessed at screening, and tumor response was assessed every 8 weeks during the induction phase, and every 12 weeks during the maintenance phase until disease progression or death (any cause) whichever occurred first, up to 9 months.
Measure: Median (Full Range); unit: Months
Arm/Group | NANT Colorectal Cancer (CRC) Vaccine
Number analyzed (Participants) | 2
Months
  RECIST | 6 [5 to 7]
  irRC | 6 [3 to 9]

4. Secondary Outcome: Duration of Response (DOR) by RECIST Version 1.1 and irRC
Description: DOR was be defined as the time from the date of first response (PR or CR) to the date of disease progression or death (any cause) whichever occurs first. Responding subjects completed study follow-up or initiating a new anticancer therapy prior to documented PD were censored in the DOR analysis at the last known date the subject was progression free prior completing follow-up or initiating the new therapy.
Time Frame: Tumors were assessed at screening, and tumor response will be assessed every 8 weeks during the induction phase, and every 12 weeks during the maintenance phase until confirmed disease progression, up to 4 months
Population: There were no participants with confirmed CR or PR. Therefore, no participants were included in the DOR analysis.
Arm/Group | NANT Colorectal Cancer (CRC) Vaccine
Number analyzed (Participants) | 0

5. Secondary Outcome: Overall Survival
Description: OS was evaluated using Kaplan-Meier methods. OS was defined as the time from the date of first treatment to the date of death (any cause). Participants who were alive at the end of follow-up were censored in the OS analysis at the last known date alive.
Time Frame: Participants were assessed from screening to death.
Measure: Median (Full Range); unit: Months
Arm/Group | NANT Colorectal Cancer (CRC) Vaccine
Number analyzed (Participants) | 2
Months | 8 [7 to 9]

6. Secondary Outcome: Disease Control Rate (Confirmed Complete Response, Partial Response, or Stable Disease Lasting for at Least 2 Months) by RECIST Version 1.1.
Description: Disease control is defined as subjects with a confirmed CR, PR, or SD lasting for at least 2 months.
Time Frame: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | NANT Colorectal Cancer (CRC) Vaccine
Number analyzed (Participants) | 2
Participants
  Confirmed CR | 0
  Confirmed PR | 0
  Stable Disease | 2
  Progressive Disease | 0

7. Secondary Outcome: Quality of Life by Patient Reported Outcomes (PRO)
Description: PROs were assessed using the Functional Assessment of Cancer Therapy-colorectal cancer (FACT-C) questionnaire. The FACT-Hep is compilation of general questions divided into five QOL subscales:
  Physical Well-Being - Scores ranging from 0-28 Social/Family Well-Being - Scores ranging from 0-28 Emotional Well-Being - Scores ranging from 0-24 Functional Well-Being - Scores ranging from 0-28 Additional Concerns - Scores ranging from 0-36 It uses 5-point Likert-type response categories ranging from 0 = 'not at all' to 4 = 'very much' The higher scales and subscales indicate better quality of life. Negatively worded items were reverse scored. If the missing for each subscale was less than 50%, the prorating scores were computed for the subscale.
Time Frame: Assessments occurred at Baseline, Cycle 2 Day 8 (C2D8), Cycle 5 Day 1 (C5D1), at an unscheduled visit prior to end of treatment, and at end of treatment (up to 5 months). Each cycle was 28 days.
Population: The questionnaire was not completed for every patient at every visit.
Measure: Median (Full Range); unit: score on a scale
Arm/Group | NANT Colorectal Cancer (CRC) Vaccine
Number analyzed (Participants) | 2
score on a scale
  Physical Well-Being - Baseline | 19 [11 to 27]
  Physical Well-Being - C2D8: number analyzed (Participants) | 1
  Physical Well-Being - C2D8 | 24 [24 to 24]
  Physical Well-Being - C5D1: number analyzed (Participants) | 1
  Physical Well-Being - C5D1 | 17 [17 to 17]
  Physical Well-Being - Unscheduled: number analyzed (Participants) | 1
  Physical Well-Being - Unscheduled | 5 [5 to 5]
  Physical Well-Being - End of treatment | 13 [7 to 19]
  Social/Family Well-Being - Baseline | 21 [19 to 22]
  Social/Family Well-Being - C2D8: number analyzed (Participants) | 1
  Social/Family Well-Being - C2D8 | 15 [15 to 15]
  Social/Family Well-Being - C5D1: number analyzed (Participants) | 1
  Social/Family Well-Being - C5D1 | 16 [16 to 16]
  Social/Family Well-Being - Unscheduled: number analyzed (Participants) | 1
  Social/Family Well-Being - Unscheduled | 17 [17 to 17]
  Social/Family Well-Being - End of treatment | 19 [15 to 22]
  Emotional Well-Being - Baseline | 19 [18 to 20]
  Emotional Well-Being - C2D8: number analyzed (Participants) | 1
  Emotional Well-Being - C2D8 | 18 [18 to 18]
  Emotional Well-Being - C5D1: number analyzed (Participants) | 1
  Emotional Well-Being - C5D1 | 21 [21 to 21]
  Emotional Well-Being - Unscheduled: number analyzed (Participants) | 1
  Emotional Well-Being - Unscheduled | 13 [13 to 13]
  Emotional Well-Being - End of treatment | 17 [17 to 17]
  Functional Well-Being - Baseline | 17 [13 to 21]
  Functional Well-Being - C2D8: number analyzed (Participants) | 1
  Functional Well-Being - C2D8 | 18 [18 to 18]
  Functional Well-Being - C5D1: number analyzed (Participants) | 1
  Functional Well-Being - C5D1 | 14 [14 to 14]
  Functional Well-Being - Unscheduled: number analyzed (Participants) | 1
  Functional Well-Being - Unscheduled | 5 [5 to 5]
  Functional Well-Being - End of treatment | 9 [8 to 9]
  Additional Concerns - Baseline | 24 [16 to 32]
  Additional Concerns - C2D8: number analyzed (Participants) | 1
  Additional Concerns - C2D8 | 28 [28 to 28]
  Additional Concerns - C5D1: number analyzed (Participants) | 1
  Additional Concerns - C5D1 | 29 [29 to 29]
  Additional Concerns - Unscheduled: number analyzed (Participants) | 1
  Additional Concerns - Unscheduled | 14 [14 to 14]
  Additional Concerns - End of treatment | 23 [14 to 31]

8. Secondary Outcome: Disease Control Rate (Confirmed Complete Response, Partial Response, or Stable Disease Lasting for at Least 2 Months) by irRC
Description: Disease control is defined as subjects with a confirmed CR, PR, or SD lasting for at least 2 months.
Time Frame: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | NANT Colorectal Cancer (CRC) Vaccine
Number analyzed (Participants) | 2
Participants
  irCR | 0
  irPR | 0
  irSD | 2
  irPD | 0

ADVERSE EVENTS:
Time Frame: Non-serious AEs were followed for 30 days after the subject's last dose of study treatment, up to 6 months. Non-serious grade 3 or 4 AEs were followed until resolution or stabilization, up to 6 months. All SAEs that had not resolved upon discontinuation of the subject's participation in the study were followed until recovered, recovered with sequelae, not recovered (death due to other cause), death (due to the SAE), lost to follow-up, up to 6 months.
Description: The numbers of participants at risk for Serious Adverse Events, All-Cause Mortality and Other (Not Including Serious) Adverse Events are zero in Regorafenib group because there are no subjects enrolled in Regorafenib group.
Arm/Group | NANT Colorectal Cancer (CRC) Vaccine | Regorafenib
All-Cause Mortality (participants affected / at risk) | 2/2 | 0/0
Serious Adverse Events (participants affected / at risk) | 1/2 | 0/0
Other Adverse Events (participants affected / at risk) | 2/2 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | NANT Colorectal Cancer (CRC) Vaccine (N=2) | Regorafenib (N=0)
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | NANT Colorectal Cancer (CRC) Vaccine (N=2) | Regorafenib (N=0)
Anaemia (Blood and lymphatic system disorders) | 2 | 0
Neutropenia (Blood and lymphatic system disorders) | 2 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0
Vision blurred (Eye disorders) | 2 | 0
Nausea (Gastrointestinal disorders) | 2 | 0
Stomatitis (Gastrointestinal disorders) | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Chills (General disorders) | 2 | 0
Fatigue (General disorders) | 2 | 0
Injection site reaction (General disorders) | 2 | 0
Pyrexia (General disorders) | 2 | 0
Pain (General disorders) | 1 | 0
Candida infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 2 | 0
Weight decreased (Investigations) | 2 | 0
Blood creatinine increased (Investigations) | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 0
Tachycardia (Cardiac disorders) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung opacity (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-28): https://cdn.clinicaltrials.gov/large-docs/57/NCT03563157/Prot_SAP_000.pdf